CLINICAL TRIAL: NCT00506324
Title: Oropharyngeal Function After Radiotherapy With IMRT
Status: Terminated | Type: Observational
Why Stopped: Physician deceased
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DC007659-01A1 (NIH); R01DC007659 (NIH)
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Head and Neck Neoplasms
Keywords: Intensity Modulated Radiotherapy; Chemotherapy; Head and Neck Neoplasms; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project defines the effect on swallowing of intensity modulation during radiotherapy in an organ preservation treatment involving chemoradiation for 125 oral, laryngeal, and pharyngeal cancer patients with previously untreated Stage III or IV disease and to identify optimum treatment strategies. The specific aims are: 1) define the physiologic effects of chemoradiotherapy with IMRT to various sites in the upper aerodigestive/vocal tract including the cervical esophagus and the rate at which patients return to oral intake; 2) document the acute toxicities, late complications, locoregional failure and survival, and the relationship between fibrosis rating and the measure of laryngeal elevation; 3) determine whether the patient's swallowing mechanism can compensate for physiologic deficits in swallowing by introduction of interventions (postural changes, voluntary swallow maneuvers, several bolus volumes); 4) determine whether time to return to oral intake, effects of swallow maneuvers and/or volume, presence of an esophageal stricture and the duration of success of dilatation depends on radiation dose volume to specific structures in the head and neck; 5) define the relationship of tongue base pressure to development of esophageal stricture. Patients will be accrued from Northwestern University and University of Chicago. Effects are defined in terms of swallowing function, morbidity, toxicity and survival. Other outcome measures are the maintenance of voluntary control (flexibility) of the oropharyngeal region as indicated by the ability to correctly produce swallow maneuvers; and positive changes in cricopharyngeal opening duration with normal bolus volume shifts. Patients will be studied pretreatment, and at 1 month, 3 months, 6 months, 12 months, and 24 months post completion of chemoradiation. At each assessment, patients will receive a videofluoroscopic assessment of swallowing utilizing a standard protocol, assessment of xerostomia, mucositis, and fibrosis as well as assessment of disease status and quality of life scales. Head and neck cancer is a severe problem that affects public health. Most current treatments are a combination of radiotherapy with chemotherapy, which can result in severe swallowing problems which may make patients unwilling to accept this type of treatment. This project attempts to quantify the swallow problems associated with this specific treatment and the effects of interventions for these swallow problems.

DETAILED DESCRIPTION:
A. Subjects One hundred and twenty-five patients with disease Stages III or IV squamous cell cancers of the oral cavity, larynx or pharynx will serve as subjects.

B. Intensity Modulation and Radiotherapy Guidelines Anatomical data that is required for the planning process is acquired using a Philip's AcQSim CT simulation system. The immobilized patient is squared up relative to the bore of the Picker PQ2000S CT scanner using the ceiling and side lasers of the system. A scout view is obtained so that the superior and inferior borders of the volume study can be determined. Forty seconds prior to the commencement of image data acquisition contrast media (125 cc of Ultravist 300) is power injected at the rate of 1.3-2.0 cc/sec using a Liebel-Flarsheim device. The CT data set is acquired with 3 mm slice thickness and spacing using the spiral mode of the scanner. While the patient is on the table, the images are transferred to the VoxelQ work station that is running AcQSim software version 4.1.1. Before the patient is released a reference isocenter is established and recorded in the AcQSim system and marked on the face mask using the isocenter locating lasers of the CT simulator, if not already indicated by radio-opaque fiducials.

The physicians then outline target volumes, GTVs and CTVs, as per ICRU 50 guidelines and outline critical structures such as the brain stem, spinal cord, salivary glands, optic apparatus, etc. After this has been done, the image and structure data is transferred to either of two treatment planning work stations: the NOMOS Corvus system running software version 5.0 or the ADAC Pinnacle RTP system running software version 6.2b. A planning target margin (PTV) is added to take into account organ motion and setup uncertainty. Lateral and Anterior-Posterior digitally reconstructed radiographs (DRRs) that demonstrate the location of isocenter are produced from the AcQSim system so that correct patient positioning can be confirmed prior to the commencement of treatment.

The prescription for the target(s) defines the dose goal for the treatment, the minimal acceptable dose and percent volume that can be under dosed and the maximum acceptable dose. The prescription for radio sensitive structures sets the nominally allowed dose, the percent volume that can be overdosed, the maximum tolerable dose and the minimum dose below which no radiation damage can be observed. These specifications, for various targets and critical structures, translate into defining three points on a dose volume histogram (DVH) curve for each tissue type. The Corvus system computes the optimal beam intensity maps using a simulated annealing algorithm whereas the ADAC system uses a sequential quadratic search method to minimize a quadratic objective function, which is constructed from a set of dose-based or dose-volume-based objectives for individual regions of interest. Delivery of the dose as prescribed by the idealized maps is accomplished by using step and shoot IMRT at both institutions. In this method the beam direction incident on the patient along with field size and collimator angle is determined by the treatment planner before the software designs the IMRT intensity maps. Therefore it is important to choose beam geometries carefully so as to maximize exposure to the target and minimize exposure to critical structures as visualized in the beam's eye view. The IMRT beams are created by utilizing a standard 80 cm leaf MLC on an Elekta Sli linear accelerator.

Radiotherapy Guidelines for the proposed study:

1. All patients will have immobilization devices with treatment planning based on Computerized Tomography (CT) information in treatment position. The CT slice thickness through target will be 3mm.
2. CT and Magnetic Resonance Imaging (MRI) data will be used to define the various targets and contour normal structures. MRI information will be used when indicated. Image fusion will be used to relate CT/MRI data when necessary.
3. The field sizes and arrangements will be at the discretion of the attending Radiation Oncologist. ICRU 50 guidelines will be used for various Tumor and Target Nomenclature:

   1. The Gross Tumor Volume (GTV): All gross disease determined from clinical examination and radiographic studies.
   2. The Clinical Target Volume (CTV): The area that potentially contains microscopic disease. Lymph node groups at risk of microscopic disease will be outlined as part of corresponding CTV. The margin between each GTV and corresponding CTV can vary from 0.2cm to 2.5cm depending upon the proximity to the critical and uninvolved structures.
   3. The Planning Target Volume (PTV): Provides a margin around CTV to compensate for internal motion and set up errors. Typically a 5mm margin may be used around CTV.

Radiation Targets and Dose Specifications:

The following is the definition of targets. The radiation doses will be delivered as specified in the protocol:

1. Primary Target Volume (PTV1): Includes gross tumor volume and volume encompassing lymph nodes with moderate to high risk of metastases (first echelon nodes) and lymph nodes with low risk of metastatic disease with corresponding CTVs.
2. Secondary Target Volume (PTV2): Includes gross tumor volume and volume encompassing lymph nodes with moderate to high potential risk of metastases with corresponding CTVs.
3. Tertiary Target Volume (PTV3): Includes gross tumor volumes for the primary tumor and nodal metastases with corresponding CTVs.

Low Neck: The midjugular, low jugular, and supraclavicular nodes can be treated either with IMRT or alternatively with an AP field that is beam split to the IMRT fields. This will be at the discretion of the treating physician. If an IMRT approach is not used, then it will not be necessary to submit the DVHs for this PTV. However, if an IMRT approach is used, then it will be necessary to generate DVHs for this PTV. Radiation doses will be as in the attached protocol.

Neck Nodes: Guidelines for anatomic boundaries and CT-based delineation of neck nodes will be as per consensus Atlas on RTOG website (www.RTOG.org → Researcher → H/N Atlas).

Normal Tissues: The appropriate normal organs will be contoured. Dose Volume Histograms (DVH) will be generated. An attempt will be made to keep the maximum radiation doses to the following organs as follows; since the radiation to these structures will be at a lower fraction per day and the maximum doses to partial volumes only, we believe these are acceptable dose levels.

Brain Stem: 54 Gy Optic Nerve/Chiasm: 55 Gy Spinal Cord: 45 Gy Mandible/TM Joint: 70 Gy or 1cc of the PTV not to exceed 75 Gy Larynx 70 Gy

Parotid Glands: Attempt will be to achieve mean dose 26 Gy in at least one gland or at least 20cc of the combined volume of both parotid glands will receive 20 Gy or at least 50% of the gland will receive 30 Gy (should be achieved in at least one gland).

Toxicity Reporting:

1. For acute toxicity the NCI/CTCAE Version 3.0 will be used.
2. For late toxicity, the RTOG/EORTC late toxicity criteria will be used.

   Each treatment will be judged as being compliant with the Image guides therapy Center in St. Louis guideline as:

   1. No variation (Total Coverage): Coverage as specified in Radiation Guideline Section.

   2. Minor variation (Marginal Coverage): The 93% isodose covers between 95% to 98% of the appropriate PTV or volumes of overdose exceed those specified in Radiation Guideline Section by 5% of the PTV volume.

   3. Major variation (Miss): The 93% isodose surface covers less than 95% of the appropriate PTV or the overdose regions of the appropriate PTV are greater than 5% of the PTV volume.

   C. Data Collection Schedule Functional data will be collected on each patient at 6 points in time: pretreatment and 5 times after the completion of the chemoradiation -- 1 month, 3 months, 6 months, 12 months, and 24 months.

   1. Swallow Evaluation. At each evaluation point, each patient will receive a maximum of 33 swallows studied by videofluoroscopy with concurrent manometry.

   A 3 mm flexible catheter containing 2 solid state pressure sensors 3 cm apart will be positioned transnasally at the beginning of the study, so that one sensor is located at the base of the tongue and the second sensor is at the top of the upper esophageal sphincter. This protocol will allow the measurement of pressures generated at the tongue base. The concurrent manometry will allow us to directly measure pharyngeal pressures during swallow. All swallows will be viewed in the lateral plane except the last three 3 ml swallows viewed in the A-P plane. Subjects will not be required to swallow volumes or viscosities that they cannot manage comfortably. All such difficulties will be recorded on the data sheets.

   Videofluoroscopy Protocol (3 swallows of each combination):

   1 ml thin liquid barium 3 ml thin liquid barium 5 ml thin liquid barium 10 ml thin liquid barium 3 ml pudding

   ¼ Lorna Doone cookie with 3 ml barium paste 3 ml thin liquid barium - chin down 3 ml thin liquid barium - effortful swallow 3 ml thin liquid barium - super-supraglottic swallow 3 ml thin liquid barium - Mendelsohn maneuver 3 ml thin liquid barium - P-A view

   2. Measure of Xerostomia. At each radiographic study of swallow, the patient's stimulated saliva production will be quantified by taking the difference of the weight of a folded sterile sponge (10 x 10 cm Kerlix) before and after chewing for 2 minutes.

   3. Data Collection Regarding Onset and Nature of Oral Intake. At each of the 6 swallow data collection points, status and nature of oral and non-oral intake will also be reported, as well as the reason for non-oral intake, i.e., nausea versus swallowing disorder. The dates when the patient began to experience difficulty eating, when and why non-oral feeding began, and when partial and full oral intake began will be recorded and reported by the speech-language pathologist.

   4. Ratings of Mucositis. Oral mucositis ratings will be completed pretreatment and at the same 5 intervals after treatment. The scale rates ulceration on a 4-point scale (0 = no lesions to 3 = a lesion > 3 cm2) and erythema on a 3-point scale (0 = none; 1 = not severe; 2 = severe) at 10 locations in the oral cavity (upper and lower lip, right and left cheek, right and left ventral and lateral tongue, floor of mouth, soft palate/fauces and hard palate). The mucositis ratings will be done by the participating speech-language pathologist (SLP) trained in using the scale.

   5. Patient's Perception of Function. A data form has been developed to define the patient's perception of swallowing function, as well as dry mouth. The patient completes the four-page form himself.

   6. QOL scales: Performance Status Scale for Head and Neck Cancer (PSS-HN) (List et al., 1990): This brief 3-part questionnaire will be given by the SLP at each evaluation point; The M.D. Anderson Dysphagia Inventory (MDADI) is a 20-item self-administered scale that investigates the impact of dysphagia on the patient's quality of life; The University of Washington Quality of Life scale (UW QOL) is a 6 item clinician-administered scale.

   7. Survival and Locoregional failure: Patients will be followed for overall survival, relapse free survival and locoregional failure. The locoregional failure pattern will be categorized as within a) Primary Target Region (PTV1); b) Secondary Target Region (PTV2) or c) Tertiary Target Region (PTV3).

ELIGIBILITY:
Inclusion Criteria:

* The target population for this study is 125 patients with stages III or IV squamous cell lesions of the oral cavity, oropharynx, pharynx or larynx, or unknown primary.

Exclusion Criteria:

* No patient will have had prior treatment for head and neck cancer or any otolaryngologic or neurologic disorder affecting swallow and no preexisting swallowing disorder.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and twenty-five patients with disease Stages III or IV squamous cell cancers of the oral cavity, larynx or pharynx will serve as subjects. No patient will have had prior treatment for head and neck cancer or any otolaryngologic or neurologic disorder affecting swallow, and no preexisting swallowing disorder.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2006-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
percent oral intake | 12 months post-treatment completion
  The percent of nutrition taken by mouth

SECONDARY OUTCOMES:
normal diet | 12 months post-treatment completion
  The patient has a normal diet when he or she includes all consistencies (thin liquid, thick liquid, pudding, pureed, soft mechanical, hard mechanical)

CONTACTS AND LOCATIONS:
Overall Officials: Jerilyn Logemann, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States